CLINICAL TRIAL: NCT06187506
Title: A Prospective, Open, Single-center Clinical Study of Disitamab Vedotin Combined With BCG Therapy in HER2-expressing High-risk Non-muscle Invasive Bladder Cancer
Brief Title: Disitamab Vedotin Combined With BCG Therapy in HER2-expressing High-risk Non-muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48C066
Record Dates: First submitted 2023-12-13; First posted 2024-01-02 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Non-muscle Invasive Bladder Cancer; HER-2 Protein Overexpression
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — disitamab vedotin; BCG Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48+BCG (Experimental): Disitamab Vedotin (2.0 mg/kg, administered intravenously every three weeks); BCG therapy: Induction therapy, i.e., intravesical therapy once a week for 6 weeks. maintenance therapy, i.e., one course of maintenance therapy at three, six and twelve months after surgery, each course once a week for 3 weeks.
  Interventions: Drug: Disitamab vedotin; Drug: Bacillus Calmette Guerin Vaccine

INTERVENTIONS:
Drug: Disitamab vedotin — 2.0 mg/kg, administered intravenously every three weeks
  Other Names: RC48
Drug: Bacillus Calmette Guerin Vaccine — Induction therapy, i.e., intravesical therapy once a week for 6 weeks. maintenance therapy, i.e., one course of maintenance therapy at three, six and twelve months after surgery, each course once a week for 3 weeks.
  Other Names: BCG

SUMMARY:
This is a prospective, open, single-center clinical study of the anti-HER2(Human epidermal growth factor receptor-2) ADC(antibody-drug conjugate) drug Disitamab Vedotin in combination with BCG(bacillus Calmette-Guerin) therapy in very high-risk NMIBC(Non-muscle invasive bladder cancer) patients with HER2 expression (IHC 1+/2+/3+), which is being conducted in accordance with the Good Clinical Practice for Pharmaceutical Trials (GCP). Approximately 20 subjects will be enrolled in this study to evaluate the efficacy and safety of Disitamab Vedotin (2.0 mg/kg, administered intravenously every three weeks) in combination with BCG therapy.

DETAILED DESCRIPTION:
The study will include patients with very high risk NMIBC with HER2 expression (IHC 1+/2+/3+) who refuse to undergo cystectomy or do not meet the requirements for cystectomy. Reasons for unsuitability or refusal of cystectomy will be documented on an electronic case report form (eCRF).

Subjects will receive 6 months of Disitamab Vedotin therapy and at least 1 year of BCG therapy. EFS(Event free survival) and CR(Complete response) rates will be evaluated after treatment by cystoscopy, pathologic histology, urine cytology, laboratory tests, and imaging. Cystoscopy and urine cytology every three months for two years, and radiography every six months. Cystoscopy and urine cytology were done every six months and radiography once a year after two years.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Histologically confirmed non-muscle-invasive urothelial cell carcinoma (UCC) of the bladder; A.Histopathology: any variant of UCC, The presence of any lymphovascular infiltration (LVI) was considered evidence of high risk. B. Confined to the mucosal (Ta, Tis) and lamina propria layers (T1) of the bladder. In addition, subjects had all visible tumors removed as completely as possible prior to the first dose of study drug and documented at baseline cystoscopy. C. CIS(Carcinoma in situ) does not require complete resection, but coexisting papillary carcinoma must be removed as completely as possible prior to enrollment and documented at baseline cystoscopy. Negative urine cytology results against malignant tumor cells are not required.
3. Presence of HER2 expression (IHC 1+/2+/3+) by IHC in our pathology department;
4. VHR(Very high risk) NMIBC, defined as having at least 1 of the following: Multiple and/or large (greater than [>] 3 centimeters [cm]) T1, (HG/G3) tumors; T1, (HG/G3) tumor with concurrent CIS; T1, G3 with CIS in prostatic urethra; Micropapillary variant of non-muscle invasive urothelial carcinoma;
5. Received first dose of medication ≤ 12 weeks from first TURBT;
6. Refusal or unsuitability for radical cystectomy;
7. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (</=) 1;
8. Adequate hematologic and end-organ function, Creatinine clearance >/=30 milliliters per minute (mL/min) (calculated using the Cockcroft-Gault formula);
9. Subjects (or their legal representatives) must sign an informed consent form (ICF);
10. Females of childbearing potential must have a negative pregnancy test result (beta-hCG) (urine or serum) within 7 days prior to the first dose of study drug.

Exclusion Criteria:

1. Evidence of locally advanced, metastatic, muscle-invasive, and/or extravesical bladder cancer;
2. Upper urinary tract urothelial carcinoma(UTIC), except 2 years without recurrence after previous radical UTUC;
3. Histopathologic examination reveals any small cell component of the bladder, simple adenocarcinoma, simple squamous cell carcinoma or simple squamous CIS;
4. Previously received other anti-HER-2 therapy;
5. Active malignancy outside of the disease being treated by the study (i.e., disease progression or need for change in therapy within the past 24 months);Only the following special cases are allowed: a. Skin cancer treated within the last 24 months and completely cured; b. Adequately treated lobular carcinoma in situ (LCIS) and ductal CIS; c. History of localized breast cancer and receiving anti-hormonal drugs or history of localized prostate cancer (N0M0) and receiving androgen blockade therapy.
6. History of uncontrolled cardiovascular disease, Included: 1) presence of any of the following in the past 3 months: unstable angina, myocardial infarction, ventricular fibrillation, torsional ventricular tachycardia, cardiac arrest or known congestive New York Heart Association class III-IV heart failure, cerebrovascular accident, or transient ischemic attack. 2) Prolonged QTc intervals confirmed by ECG evaluation during screening(Fridericia; QTc>480 ms). 3) Pulmonary embolism or other venous thromboembolism within the past 2 months.
7. Pregnant or lactating women;
8. Known infection with human immunodeficiency virus (HIV), unless the subject has been on stable antiretroviral therapy for the past 6 months or longer and has not had an opportunistic infection in the past 6 months and has had a CD4 count >350 in the past 6 months;
9. Evidence of active hepatitis B or C infection (e.g., subjects with hepatitis B who have a history of hepatitis C but have a normal polymerase chain reaction test result for hepatitis C virus and who are positive for antibodies to hepatitis B surface antigen may be enrolled in the study);
10. Have not recovered from toxic effects of previous anticancer therapy (except for toxic effects of no clinical significance, such as alopecia, skin discoloration, neuropathy and hearing impairment).
11. Delayed wound healing, defined as skin/decubitus ulcers, chronic leg ulcers, known gastric ulcers, or non-healing incisions;
12. Major surgery within 4 weeks prior to day 1 of cycle 1 (TURBT not considered major surgery);
13. Other patients assessed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With CR as Assessed by the Investigator according to Cystoscopy and Urine Cytology at Month 3 | up to 3 months
  CR at the 3-month disease assessment, evaluated by both cystoscopy and cytology.
Event-Free Survival (EFS) rate, as Assessed according to Cystoscopy and Urine Cytology | up to 6 months
  Percentage of Participants With Event-Free Survival (EFS), as assessed according to Cystoscopy and Urine Cytology ( patients who are alive and free of persistent/recurrent high-grade NMIBC.)

SECONDARY OUTCOMES:
Percentage of Participants With CR as Assessed by the Investigator according to Cystoscopy and Urine Cytology at Month 6, 12 | up to 12 months from the date of randomization as assessed by the investigator according to cystoscopic assessment and urine cytology
  CR at the 6, 12-month disease assessment, evaluated by both cystoscopy and cytology.
Duration of CR will be defined for participants with a CR as the time from the first occurrence of a documented complete response to recurrence of high-grade NMIBC or death from any cause. | From first occurence of a documented CR until the time of recurrence of NMIBC or death from any cause, whichever came first, assessed up to 24 months
  Duration of CR will be defined for participants with a CR as the time from the first occurrence of a documented complete response to recurrence of high-grade NMIBC or death from any cause.
Percentage of Participants With Event-Free Survival (EFS), as Assessed according to Cystoscopy and Urine Cytology | up to 24 months
  EFS rate at 12, 24 months, defined as the proportion of patients who are alive and free of persistent/recurrent high-grade NMIBC.
Progression-Free Survival (PFS), as Assessed according to Cystoscopy and Urine Cytology | Time from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  PFS, defined as the time from the first study treatment to the first occurrence of progression to muscle-invasive disease based on cystoscopy and urine cytology or death from any cause.
Overall Survival | Time from date of randomization to death from any cause, assessed up to 60 months
  defined as the time from first study treatment to death from any cause
Percentage of Participants With Adverse Events | up to 24 months
  Percentage of participants with at least one adverse event during the study

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No